CLINICAL TRIAL: NCT01558557
Title: Gluten Free Diet in People With Schizophrenia: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, MPRC, Deanna L. Kelly, Pharm.D., BCPP, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00041292
Record Dates: First submitted 2012-03-15; First posted 2012-03-20 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Gluten Sensitivity; Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gluten Free Diet (Experimental)
  Interventions: Other: Gluten Free Diet

INTERVENTIONS:
Other: Gluten Free Diet — Participants will be given a Gluten Free Diet for 2 weeks

SUMMARY:
Background: Celiac disease is an immune-mediated reaction to gluten, presenting with diarrhea, weight loss, abdominal complaints and a range of less common associated neurologic and psychiatric symptoms. Evidence of a link between schizophrenia and celiac disease dates back to 1961. Recent evidence shows that 5.5% (age adjusted) of persons with schizophrenia participating in the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) study had a level of antibodies to tTG that is consistent with a diagnosis of celiac disease (compared to 1.1% of the comparison sample). An unexpected finding was that 23.4% (age adjusted) of the CATIE sample had antibodies to gliadin (compared to 2.9% of the comparison sample). It is hypothesized that a gluten free diet in people with schizophrenia who have Celiac disease or gluten sensitivity will have improvement in symptoms and quality of life.

Objectives: The aim of this proposed pilot study is to establish the feasibility of a initiating and maintaining a Gluten-free diet in these two groups. For this study The investigators will identify 8 individuals who have positive assays to tTG antibodies and confirmed celiac disease (N=4), or positive assays for anti-gliadin antibodies (N=4). The investigators plan to consent at least 2 subjects from each group and ask them to participate in a two-week open label treatment of a gluten free diet. The groups are;

1. Celiac disease (positive tTG antibody); and
2. Positive assay on Antigliadin antibodies

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be of either gender and of any race, with an age range of 18 55.
* Subjects will meet DSM-IV (APA, 1994) criteria for either schizophrenia or schizoaffective disorder. A best estimate diagnostic approach will be utilized in which information from the Structured Clinical Interview for DSM-IV (First et al, 1997) is supplemented by information from family informants, previous psychiatrists, and medical records to generate a diagnosis.
* Subjects will be required to have celiac disease (positive tTG antibody) or have gluten sensitivity (positive or AGA antibodies).
* Must be clinically stable and on the same antipsychotic for at least two months with an unchanged dose for the prior four weeks.
* Participants must complete the Evaluation to Sign Consent with a score of 10/12 or higher.

Exclusion Criteria:

* Pregnant or lactating women will be excluded. Pregnancy will be determined by pregnancy test. Lactating will be determined by participant report.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2008-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in symptoms from baseline to end of study | Baseline and 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, Pharm.D., BCPP, Principal Investigator — Principal Investigator
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States